CLINICAL TRIAL: NCT01596569
Title: Combining Cognitive Treatment With Noninvasive Brain Stimulation in Blast TBI
Brief Title: Combined Transcranial Magnetic Stimulation and Cognitive Treatment in Blast Traumatic Brain Injury
Acronym: COST-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Yelena Bogdanova, PhD, BUMC Faculty, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: H-29706; UL1RR025771 (NIH)
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Brain Injury; Cognitive Dysfunction; Blast Injury
Keywords: Blast Traumatic Brain Injury; Cognitive Rehabilitation; Transcranial Magnetic Stimulation; Combined Treatment
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction; Blast Injuries | interventions — Transcranial Magnetic Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TMS and Cognitive Intervention (Active Comparator): Active TMS and Cognitive Intervention:
  Repetitive Transcranial Magnetic Stimulation (rTMS) and Cognitive intervention designed specifically to address the most common cognitive deficits (executive function and memory).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Cognitive Intervention
- Sham TMS and Cognitive Intervention: (Sham Comparator): Sham TMS and Cognitive Intervention:
  Repetitive Transcranial Magnetic Stimulation (rTMS) and Cognitive intervention designed specifically to address the most common cognitive deficits (executive function and memory).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Cognitive Intervention

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Daily rTMS treatment for one week. Sham TMS participants receive the same study procedures as patients receiving active TMS.
  Other Names: Transcranial Magnetic Stimulation; Noninvasive Brain Stimulation; Magstim Corporation
Behavioral: Cognitive Intervention — Cognitive intervention designed specifically to address the most common cognitive deficits (executive function and memory) in bTBI.
  All participants receive weekly cognitive treatment sessions for 10 weeks.
  Other Names: Cognitive Rehabilitation; Cognitive Training

SUMMARY:
This study investigates the efficacy of a novel neurorehabilitation program combining noninvasive brain stimulation (transcranial magnetic stimulation or TMS) and cognitive therapy, on cognitive function and quality of life in individuals with blast-induced traumatic brain injury (bTBI).

DETAILED DESCRIPTION:
The most common blast-induced traumatic brain injury (bTBI)-associated problems are cognitive deficits, such as executive functioning and memory. This study evaluates a combined rehabilitation program: transcranial magnetic stimulation (TMS) and cognitive therapy for treatment of patients with bTBI. TMS is a noninvasive way of stimulating the brain, which is not painful and does not involve any needles or any form of surgery. It acts by delivering a magnetic stimulation to a particular brain region. Half of the study participants will receive cognitive intervention with active TMS, and a control group will receive cognitive intervention with sham TMS. This study takes place in Boston, Massachusetts: at the VA Boston Healthcare System and Beth Israel Deaconess Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF active-duty personnel or veterans exposed to blast
* Meets criteria for mild TBI
* LOC of 30 min or less
* Age: 21-50
* Primary language is English

Exclusion Criteria:

* Evidence of penetrating head injury
* History of previous neurological diagnosis
* History of previous psychotic disorder prior to the blast exposure
* Hearing or vision impairment

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-11-18 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
Post concussive symptoms in TBI | 4 weeks
  Neurobehavioral Symptoms Inventory (NSI) is a 22-item measure that assesses the post-concussive symptoms in patients with TBI.The NSI asks the patient to rate each of the symptoms according to how much the symptom has disturbed him/her using a five point scale. Patient ratings are based on descriptions of the frequency of the symptom, the extent to which the symptom disrupts the patient's activities, and the patient's perceived need for help with the symptom. A total score will be summated. Lower scores are more favorable.

SECONDARY OUTCOMES:
Daily life and functional outcome | 4 weeks
  Dysexecutive Questionnaire (DEX) is a 20-item self-report measure of real-life deficits relevant to cognitive/executive function that measures four domains: emotional, motivational, behavioral and cognitive. All items are rates in terms of frequency on a 5-point scale: 0 (never), 1(occasionally), 2 (sometimes), 3 (fairly often), 4 (very often). Scores are summed and the total scores range from 0 to 80, with higher scores indicating greater problems with executive functioning.
PTSD symptoms | 4 weeks
  Military version (PCL-M) 17-item self-report measure that assesses PTSD symptoms. Each item is scored on the frequency of the problem from 1 to 5 where 1= not at all and 5= extremely. A total score is calculated and lower scores are more favorable..

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Bogdanova, PhD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - VA Boston Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogdanova Y, Verfaellie M. Cognitive sequelae of blast-induced traumatic brain injury: recovery and rehabilitation. Neuropsychol Rev. 2012 Mar;22(1):4-20. doi: 10.1007/s11065-012-9192-3. Epub 2012 Feb 17. PMID 22350691